CLINICAL TRIAL: NCT03571776
Title: Anti-mullerian Hormone in Ovarian Reserve Evaluation After Treatment of Endometriomas With Alcohol Sclerotherapy Versus Surgery: Clinical Trial
Brief Title: Anti-mullerian Hormone (AMH) After Treatment of Endometriomas With Alcohol Sclerotherapy Versus Surgery: Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment because patients and gynecologists prefer the sclerosis arm to avoid surgery
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Amparo Garcia-Tejedor, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR031/18
Record Dates: First submitted 2018-05-31; First posted 2018-06-28 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Endometrioma; Fertility Disorders
MeSH Terms: conditions — Endometriosis | interventions — Surgical Procedures, Operative; Sclerotherapy

STUDY DESIGN:
Intervention Model Description: Multicenter, National, assignment 1: 1, stratified by age, previous oophorectomy and uni- or bilateral ovarian involvement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Active Comparator): Laparoscopic ovarian cystectomy
  Interventions: Procedure: Surgery
- Sclerotherapy (Active Comparator): US-aspiration and alcohol sclerosis
  Interventions: Procedure: Sclerotherapy

INTERVENTIONS:
Procedure: Surgery — Laparoscopic ovarian cystectomy
  Arms: Surgery
Procedure: Sclerotherapy — US-aspiration and alcohol sclerosis
  Arms: Sclerotherapy

SUMMARY:
The purpose of this multicenter study is to compare the ovarian reserve after alcohol sclerosis of the endometriomas against conventional surgery (AMH, follicle stimulating hormone (FSH) and antral follicles count) as well as the complications and costs between the 2 procedures.

DETAILED DESCRIPTION:
Clinical Trial Phase III, Multicenter, National, open, parallel-group assignment 1: 1, stratified by age, previous oophorectomy and uni- or bilateral ovarian involvement. Patients with suspected ovarian endometrioma by ultrasound will be randomized into 2 groups: (a) Study Group: echoguided aspiration plus sclerosis with alcohol; (B) Control group: Laparoscopic Cystectomy. Pre-treatment, and 6 months after treatment, AMH values will be determined. Complications, recurrences and costs from each treatment will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilocular endometrioma according ultrasounds
* Endometrioma size: 30-100 mm when symptoms were present and 50-100 mm if asymptomatics
* > 3 months from diagnosis
* Ca125 <200 IU/mL and human epididymis protein 4 (HE4) < 70,

Exclusion Criteria:

* Previous gynecological cancer
* Symptomatic severe extraovarian endometriosis
* Dermoid or high risk of malignancy cysts
* Pregnancy
* Mental disability

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline AMH Test | prior and 6 months after both procedures
  the value of AMH in ng/mL

SECONDARY OUTCOMES:
Change from Baseline antral follicles count | prior and 6 months after both procedures
  US antral follicles count
Complications | 1 month after the procedure
  number of participants with complications
Costs | 1 month after the procedure
  costs (euros) of the procedure plus cost of their complications
Change from Baseline Pain | prior and 6 months after both procedures
  Visual Analog Score for pain (ranged 1-10). Patients pain evaluation fron 1 no pain to 10 maximum pain considered

CONTACTS AND LOCATIONS:
Overall Officials: Amparo Garcia-Tejedor, MDPhD, Principal Investigator — Hospital de Bellvitge. IDIBELL
Locations (1):
- Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coccia ME, Rizzello F, Cammilli F, Bracco GL, Scarselli G. Endometriosis and infertility Surgery and ART: An integrated approach for successful management. Eur J Obstet Gynecol Reprod Biol. 2008 May;138(1):54-9. doi: 10.1016/j.ejogrb.2007.11.010. Epub 2008 Feb 20. PMID 18243485
- [Background] Muzii L, Bianchi A, Croce C, Manci N, Panici PB. Laparoscopic excision of ovarian cysts: is the stripping technique a tissue-sparing procedure? Fertil Steril. 2002 Mar;77(3):609-14. doi: 10.1016/s0015-0282(01)03203-4. PMID 11872220
- [Background] Akamatsu N, Hirai T, Masaoka H, Sekiba K, Fujita T. [Ultrasonically guided puncture of endometrial cysts--aspiration of contents and infusion of ethanol]. Nihon Sanka Fujinka Gakkai Zasshi. 1988 Feb;40(2):187-91. Japanese. PMID 3283269
- [Background] Noma J, Yoshida N. Efficacy of ethanol sclerotherapy for ovarian endometriomas. Int J Gynaecol Obstet. 2001 Jan;72(1):35-9. doi: 10.1016/s0020-7292(00)00307-6. PMID 11146075
- [Background] Kafali H, Eser A, Duvan CI, Keskin E, Onaran YA. Recurrence of ovarian cyst after sclerotherapy. Minerva Ginecol. 2011 Feb;63(1):19-24. PMID 21311417
- [Result] Raffi F, Metwally M, Amer S. The impact of excision of ovarian endometrioma on ovarian reserve: a systematic review and meta-analysis. J Clin Endocrinol Metab. 2012 Sep;97(9):3146-54. doi: 10.1210/jc.2012-1558. Epub 2012 Jun 20. PMID 22723324
- [Result] Biacchiardi CP, Piane LD, Camanni M, Deltetto F, Delpiano EM, Marchino GL, Gennarelli G, Revelli A. Laparoscopic stripping of endometriomas negatively affects ovarian follicular reserve even if performed by experienced surgeons. Reprod Biomed Online. 2011 Dec;23(6):740-6. doi: 10.1016/j.rbmo.2011.07.014. Epub 2011 Jul 27. PMID 22019621
- [Result] Yazbeck C, Madelenat P, Ayel JP, Jacquesson L, Bontoux LM, Solal P, Hazout A. Ethanol sclerotherapy: a treatment option for ovarian endometriomas before ovarian stimulation. Reprod Biomed Online. 2009 Jul;19(1):121-5. doi: 10.1016/s1472-6483(10)60055-7. PMID 19573300
- [Result] Garcia-Tejedor A, Castellarnau M, Ponce J, Fernandez ME, Burdio F. Ethanol sclerotherapy of ovarian endometrioma: a safe and effective minimal invasive procedure. Preliminary results. Eur J Obstet Gynecol Reprod Biol. 2015 Apr;187:25-9. doi: 10.1016/j.ejogrb.2015.02.004. Epub 2015 Feb 16. PMID 25739052
- [Result] Somigliana E, Berlanda N, Benaglia L, Vigano P, Vercellini P, Fedele L. Surgical excision of endometriomas and ovarian reserve: a systematic review on serum antimullerian hormone level modifications. Fertil Steril. 2012 Dec;98(6):1531-8. doi: 10.1016/j.fertnstert.2012.08.009. Epub 2012 Sep 10. PMID 22975114
- [Derived] Garcia-Tejedor A, Guevara-Peralta R, Martinez-Garcia JM, Corbalan S, Aguero M, Gomez-Romero M, Cararach M, Castellarnau M, Rodriguez M, Lou-Mercade AC, Costa L, Rodriguez MJ, Huguet E, Carreras M, Castel-Segui AB, Font-Roig M, Royo S, Sarasa N, Candas B, Perez-Carton S, Ortega C, Pla MJ, Ponce J. Ultrasound-guided ethanol sclerotherapy versus laparoscopic surgery for endometriomas: a randomized clinical trial in a real-world setting. Arch Gynecol Obstet. 2025 Dec;312(6):2199-2210. doi: 10.1007/s00404-025-08205-1. Epub 2025 Nov 4. PMID 41186685